CLINICAL TRIAL: NCT04949568
Title: Self-Management and Glycemic Control in Adult Haitian Immigrants With Type 2 Diabetes: A Pilot Randomized Study
Brief Title: Self-Management and Glycemic Control in Adult Haitian Immigrants With Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-9103
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2; Patient Engagement; Patient Education
Keywords: Immigrant Health; Diabetes Mellitus, Type 2; Metabolic Diseases; Self-Management Behaviors; Haitian Americans
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Participation; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Behavioral: Diabetes Self-management behaviors
Who Masked: Participant
Masking Description: Both conditions will receive standard care. We will use sequentially numbered opaque sealed envelopes to conceal the allocation determination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetes Self-Management Behaviors (Experimental): Self-Management Education Program The culturally tailored Diabetes Self-Management Education Program involves the following: 1) an initial 45-minute face-to-face private consultation collaboratively determining goals; followed by 2) six 2-hour weekly educational interactive sessions in a format TBD by aim 1. We will deliver culturally targeted written materials and presentations in these sessions. Participants will be asked to practice self-management behaviors concurrently and for four additional weeks.
  Interventions: Behavioral: Diabetes Self-Management Behaviors
- Usual Type 2 Diabetes Care (No Intervention): The usual care arm will receive the clinic's standard type 2 diabetes care and remain under their providers' care for the duration of the study.

INTERVENTIONS:
Behavioral: Diabetes Self-Management Behaviors — The intervention is to be delivered by an interventionist.
  Arms: Diabetes Self-Management Behaviors

SUMMARY:
The objective of the study is to conduct a pilot randomized study to test feasibility and preliminary efficacy of the developed diabetes self-management education program with 40 adult Haitian immigrants.

DETAILED DESCRIPTION:
This is a two-arm randomized trial. Participants will be randomized to the culturally tailored Diabetes Self-Management Education Program or standard care condition in a 1:1 allocation. All participants will receive standard type 2 diabetes care at the enrolled clinic and remain under their providers' care for the duration of the study. The culturally tailored Diabetes Education Program involves the following: 1) an initial 45-minute face-to-face consultation; and 2) six 2-hour weekly interactive educational sessions in a format to be determined (TBD) by Aim 1 (e.g., in-person, video/telephone conference call).

ELIGIBILITY:
Inclusion Criteria:

* Self-described Haitian immigrant aged 21 and older
* Known diagnosis of type 2 diabetes for at least one year
* Have lived in the US for at least one year
* Have an HbA1c of 7.5%
* Willing and able to participate in an individual interview

Exclusion Criteria:

* Having a diagnosis of type 1 diabetes
* Unable to comprehend, consent and or fully participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Summary of Diabetes of Self-Care Activities Scale (11- item) | (T0) baseline through (T3) 90 days post-intervention
  Change in diabetes self-management behaviors (0-7, higher scores indicate improvement)
Stanford Diabetes Self-Efficacy Scale (8- item) | (T0) baseline through (T3) 90 days post-intervention
  Change in general self-efficacy 1-10, higher scores indicate improvement)
Wrist-worn actigraphy (ActiGraph) to be worn while awake | (T0) baseline through (T3) 90 days post-intervention
  Change in physical activity (Frequent physical activity indicates improvement)
Glucose Variability data from continuous glucose monitor (CGM) will be downloaded directly from participants provided (blinded) FreeStyle Libre Pro | (T0) baseline through (T3) 90 days post-intervention
  Time in range and glucose variability (More time in range and less glucose variability indicates improvement)

SECONDARY OUTCOMES:
Diabetes Distress Scale (DDS) (17-item), using Numerical Rating Scale: 0-6 | (T0) baseline through (T3) 90 days post-intervention
  Change in diabetes distress ( 0-6, lower scores indicates improvement)

CONTACTS AND LOCATIONS:
Overall Officials: Cherlie Magny-Normilus, PhD, FNP-BC, FAAN, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magny-Normilus C, Whittemore R, Wexler DJ, Schnipper JL, Nunez-Smith M, Fu MR. Barriers to Type 2 Diabetes Management Among Older Adult Haitian Immigrants. Sci Diabetes Self Manag Care. 2021 Oct;47(5):382-390. doi: 10.1177/26350106211040435. PMID 34610761